CLINICAL TRIAL: NCT02371330
Title: The Neonatal Hemorrhagic Risk Assessment in Thrombocytopenia Study - Neo-HAT Study
Brief Title: The Neonatal Hemorrhagic Risk Assessment in Thrombocytopenia Study
Acronym: Neo-HAT
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Emoke Deschmann, M.D., M.M.Sc., Attending Neonatologist, Karolinska Institutet
Other Study IDs: TRF-1516
Record Dates: First submitted 2015-02-13; First posted 2015-02-25 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Thrombocytopenia
Keywords: Thrombocytopenia; Neonate; PFA-100; Neo-BAT; Hemorrhage
MeSH Terms: conditions — Thrombocytopenia; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This is a prospective longitudinal study that evaluates Platelet Function Analyzer-100 (PFA-100) CT-ADPs (closure time-ADP) and incidence of bleeding using the Neonatal Bleeding Assessment Tool - Neo-BAT in preterm neonates <32 weeks gestational age or with a birth weight <1500 grams and with different degrees of thrombocytopenia.

The investigators hypothesized that PFA-100 CT-ADP, a global in vitro test of primary hemostasis, will be a better predictor of clinical bleeding in neonates than platelet count alone. A bleeding risk assessment marker could help physicians more accurately determine the risk/benefit ratio of platelet transfusions, guiding platelet transfusion decisions in neonates with thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

* <32 weeks gestation or with a birth weight <1500 grams;
* Have confirmed moderate-to-severe thrombocytopenia, defined as a platelet count <100x109/L;
* Have a parent/guardian willing to comply with the protocol and provide written informed consent.

Exclusion Criteria:

* Are not expected to survive by the Attending Neonatologist;
* Are thought to have a congenital thrombocytopenia or platelet dysfunction, based on family history or clinical presentation (e.g. associated congenital malformations, platelet morphology);
* Have a major chromosomal anomaly such as Trisomy 13, 18, or 21.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to the Neonatal Intensive Care Unit who are <32 weeks gestation or with a birth weight <1500 grams.
Sampling Method: Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2015-04; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Neo-BAT score (Neo-BAT: Neonatal Bleeding Assessment Tool) | study period: 5 days
  The NeoBAT is a simple, reliable and objective tool for the standardized assessment of bleeding in neonates, which was developed by an international team of experts based on the World Health Organization bleeding score for adults.

SECONDARY OUTCOMES:
Number of thrombotic events | up to post-conceptional age 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Emoke Deschmann, M.D., M.M.Sc., Principal Investigator — Department of Women's and Children's Health, Karolinska Institutet
Locations (2):
- Department of Pediatrics, Levine Children's Hospital, Carolinas Healthcare System, Charlotte, North Carolina, United States
- Astrid Lindgren Children's Hospital, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Deschmann E, Sola-Visner M, Saxonhouse MA. Primary hemostasis in neonates with thrombocytopenia. J Pediatr. 2014 Jan;164(1):167-72. doi: 10.1016/j.jpeds.2013.08.037. Epub 2013 Oct 3. PMID 24094764